CLINICAL TRIAL: NCT00921271
Title: The Application of Near Infrared Spectroscopy (NIRS) in the Detection of Lower Limb Compartment Syndrome
Status: Completed | Type: Observational
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Tom Barker, Dr, University Hospital Birmingham NHS Foundation Trust
Other Study IDs: RRK3786
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Compartment Syndrome
Keywords: Compartment syndrome
MeSH Terms: conditions — Compartment Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- At risk for compartment syndrome.: Patients admitted to Selly Oak Hospital, Birmingham, Uk, meeting one or more of the following inclusion criteria:
  1. Patients with one or more of the following injuries:
     * tibial fracture.
     * crush injury/soft tissue injury to lower limb without fracture.
     * pelvic fracture.
     * major vascular injury below the aortic bifurcation.
     * 2 or more long bone fractures.
  2. Any patient sustaining a traumatic injury with a base deficit ≥ 6 mEq/L within 12 hours of Hospital admission.
  3. Any patient receiving ≥ 6 units packed red blood cells within 12 hours of hospital admission.
  Interventions: Device: Monitoring of StO2

INTERVENTIONS:
Device: Monitoring of StO2 — Monitoring of lower limb anterior compartment StO2, taking measurements on an hourly basis for the duration of the study protocol.
  Other Names: INOVOS system.

SUMMARY:
This study aims to determine how infrared spectroscopy compares to continuous compartment pressure monitoring in the detection of compartment syndrome.

Individuals meeting the study eligibility criteria will be identified at time of admission by the receiving Trauma and Orthopaedics Registrar who will be trained in the study design and protocols.

Eligible individuals will be approached about participating in the study either at time of admission or shortly afterwards, either by the chief investigator or another doctor trained in the research protocol. Where the individual is unconscious or otherwise incapacitated, which is likely in many major trauma victims, inclusion in the study will be discussed with the patient's legal representative and/or family.

The consent process for the study will consist of having the study protocol explained by either the chief investigator, or another doctor trained in the study design. Patients will be allowed to read a participant information sheet, and permitted as much time as they require to decide if they wish to participate in the study. Verbal and written consent will be taken using a study specific consent form.

In the case of incapacitated patients, the study design will be explained to their relatives' legal representatives as appropriate and advice sought from them as to whether they know of any reason why the patient might object to participate in the study. Upon regain capacity consent will be sought from the patient for storage and analysis of their study data.

Once consented, the patient will undergo monitoring with both continuous compartment pressures, and NIRS measurements.

Recordings for both techniques will be taken each hour, as part of the patients normal observations, from the point of consent until 24 hours after their first operation. Where patients do not have an operation the total duration of monitoring will be 24 hours. The measurements will be taken by nursing staff who have received training in both techniques. The procedure for each technique is described below:

1. Continuous compartment pressures will be recorded in the broken leg, in case of tibial fractures, in all other patients fitting the inclusion criteria measurements will be taken from both legs (as both legs are at risk of compartment syndrome).

   Compartment pressures will be recorded using a slit catheter technique. Insertion of the slit catheter will be performed by either the chief investigator or Orthopaedic Registrar who will have been trained in the technique. The slit catheter is inserted using a sterile technique - the skin over the front outer part of the leg is cleaned and a catheter inserted into the anterior muscle compartment at this point. The catheter should be sited at the approximate midpoint of the leg, although this can be adjusted up or down if this would lead to insertion into a fracture site. The catheter is secured with a sterile dressing and connected to a monitor from which recordings can be taken, the catheter can be left in place for the duration of the study with no need to re-site it unless it stops recording accurately. At the same time as compartment pressure measurements are taken the patient's blood pressure will be monitored and the 'Perfusion Pressure' for the leg calculated, where:

   Perfusion pressure = diastolic blood pressure - leg compartment pressure
2. NIRS measurements will be taken with an the INVOS system, produced by Somentics. These measurements will be taken from both legs, the affected leg and other other leg used as a control for comparison. Where both legs are at risk measurements will be taken from both legs and the midpoint of the forearm used as a control.

The INVOS probe is a small adhesive patch that is stuck to the skin. The probe is sterile and will be attached using the same sterile technique as the compartment pressure catheter. Where the overlying skin is hairy the hair overlying the area for the probe should be clipped before attaching the probe, to ensure adequate adhesion and accurate readings. The probe is to be sited just below the compartment pressure catheter, although if there is an underlying haematoma (blood clot), then the probe should be positioned so at to avoid this but still remaining over the front outer part of the leg. This technique conforms with the manufacturers recommended use of the equipment and is similar protocol to previous studies.

At the end of the monitoring period both measuring devices are removed. If the patient has developed compartment syndrome during this period and required an operation, the NIRS probe and compartment pressure catheter will be replaced for a further 12 hours of monitoring to monitor the changes post-operatively and ensure compartment pressures stay low.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one or more of the following injuries:

  * tibial fracture
  * crush injury/soft tissue injury to lower limb without fracture
  * pelvic fracture
  * major vascular injury below the aortic bifurcation
  * 2 or more long bone fractures
* Any patient sustaining a traumatic injury with a base deficit ≥ 6 mEq/L within 12 hours of Hospital admission.
* Any patient receiving ≥ 6 units packed red blood cells within 12 hours of hospital admission.

Exclusion Criteria:

* Age ≤ 16 years are excluded by design, as all pediatric cases are managed at Birmingham Childrens Hospital. There is no upper age limit.
* Bilateral lower limb amputees.
* Individuals who have received methylene blue within the previous week or during the study period.
* Patient refusal to participated in the trial.
* In the case of incapacitated patients, refusal by the patient's relatives/representatives, or where no representative can be identified.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to Selly Oak Hospital (Secondary care) meeting the study inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Absolute limb StO2 at limb perfusion pressures ≤ 30 mmHg. | Hourly
Control corrected limb StO2 at limb perfusion pressures ≤ 30 mmHg. | Hourly

SECONDARY OUTCOMES:
Correlation between absolute limb StO2 and limb perfusion pressures. | Hourly
Correlation between control corrected limb StO2 and limb perfusion pressures. | Hourly
Incidence of compartment syndrome in study population. | 24 hours
Survival to discharge. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Tom Barker, MBChB, MRCS, Principal Investigator — University Hospitals Birmingham
Locations (1):
- Selly Oak Hospital, Birmingham, West Midlands, United Kingdom